CLINICAL TRIAL: NCT07343895
Title: Atrial Fibrillation and Long Term ECG Monitoring of Heart Rhythm in the Tromsø Study
Brief Title: Population-based Atrial Fibrillation Screening in Individuals With NT-proBNP Above Median in the Tromsø Study
Acronym: PAFS-Tromsø
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2025/856478 (REK)
Record Dates: First submitted 2025-07-21; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF); Stroke; NT-pro-BNP; Cognitive Function and Well-Being; Heart Failure
Keywords: ECG247; Atrial Fibrillation; Stroke; NT-Pro-BNP; Cognitive decline; Life Quality; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Heart Failure; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: In the planned open label randomized screening trial trial we plan to include 4000 individuals fra the 8th wave of the population based Tromsø Study with NT-proBNP above median without previous known AF or ongoing anticoagulant treatment. Participants will be randomized 1:1 to continuous ECG monitoring using the Norwegian produced ECG247 sensor. og to the control group without any monitoring of heart rythm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): A total of 2000 individuals with NT-proBNP levels above the median, without previously known atrial fibrillation (AF) or ongoing anticoagulation therapy, will be randomized long-term heart rhythm monitoring using ECG247 (5-7 days). Individuals with AF in the intervention group will be offered anticoagulation therapy in accordance with current guidelines.
  Interventions: Diagnostic Test: Long term heart rythm monitoring by ECG247
- Control (No Intervention): The control arm

INTERVENTIONS:
Diagnostic Test: Long term heart rythm monitoring by ECG247 — The AF screening device will be sent by post from the study centre to participants in the intervention group at inclusion, free-of-charge. User guides and a "help-desk" located at the University Hospital of North Norway will be available for phone/video assistance. Continuous ECG monitoring using the Norwegian produced ECG247 sensor will be performed for 5-7 days. Single lead ECG data is sent to a cloudbased server intermittently. The system stores information of ECG quality and is evaluated by trained algorithms which classify arrhythmias based on current criteria. All ECG recordings will be reviewed by a group of trained and experienced study nurses and physicians. In the event of clinically relevant arrhythmias, participants will be contacted as soon as possible and receive advice on follow-up with their general practitioner. Anticoagulation therapy and other treatments will be recommended if indicated according to current guidelines.
  Arms: Intervention arm

SUMMARY:
The aim is to investigate whether screening with long-term ECG monitoring in individuals with elevated NT-proBNP leads to a lower incidence of ischeamic stroke and death from vascular causes. The project is a sub-study within the 8th wave of the population based Tromsø Study. Information on previous diseases, medication use, and risk factors is collected through questionnaires, blood samples, and measurements of height, weight, blood pressure, and ECG.

A total of 4,000 individuals with NT-proBNP levels above the median, without previously known atrial fibrillation (AF) or ongoing anticoagulation therapy, will be randomized to either long-term heart rhythm monitoring (7 days) or a control group without long-term ECG monitoring (2,000 in each group). Individuals with AF in the intervention group will be offered anticoagulation therapy in accordance with current guidelines.

The intervention group and the control group will be compared with regards to incident stroke and death within a 6-year follow-up period. Information on endpoints and anticoagulation use will be obtained through linkage to national registries.

DETAILED DESCRIPTION:
This project has the potential for providing new knowledge related to the benefit of a stepwise screening approach for AF according to NT-proBNP level, utilizing a novel patch monitor with continuous ECG monitoring and automatic artificial intelligence based (AI) ECG analysis. The present project is planned as a sub-study of the epidemiological population-based Tromsø Study. In a randomized controlled clinical trial, we plan to test the primary hypothesis that in individuals with elevated NT-ProBNP who are diagnosed with AF through long-term ECG monitoring, anticoagulation treatment according to international guidelines will reduce the incidence of incident ischeamic stroke and cardiovascular death in the screening group compared to individuals who do not undergo screening (control group). The study will be performed within a well-defined cohort with extensive available longitudinal and cross-sectional information on risk factors and co-existing conditions. This setup facilitates addressing several knowledge gaps concerning risk stratification including associations between AF and echocardiographic parameters, cognitive impairment, structural changes on brain MRI, and HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years
* NT-proBNP> median level
* Informed consent for participation

Exclusion Criteria:

* History of AF (self-reported)
* Use of anticoagulation therapy
* Pacemaker/CRT device
* No available smart phone

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2032-03-01 (Estimated); Study Completion 2035-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the composite outcome of ischemic stroke or cardiovascular death | Within 6 years of screening
  Composite outcome of ischemic stroke and cardiovascular death
Number of participants with ischemic stroke | Within 6 years of screening
  Ischemic stroke outcome
Number of participants with intracerebral hemorrhage | Within 6 years of screening
  Intracerebral hemorrhage outcome
Number of participants with cardiovascular death | Within 6 years of screening
  Cardiovascular death outcome

SECONDARY OUTCOMES:
Number of participants with atrial fibrillation | Within 14 days of screening
  Atrial fibrillation prevalence
Duration of atrial fibrillation in hours | Within 14 days of screening
  Atrial fibrillation burden
Left atrial volume index | Within 1 year of screening
  Echocardiographic measure
Left atrial reservoir strain | Within 1 year of screening
  Echocardiographic measures
Score on the 12-word immediate recall test | Within 6 years of screening
  Cognitive test performance outcome
Score on the Mini-Mental State Examination (MMS-E) | Within 6 years of screening
  Cognitive test performance outcome
Score on the digit symbol coding test | Within 6 years of screening
  Cognitive test performance outcome
Score on the HRQoL EuroQol-5 Dimension (EQ5D) | Within one year of screening
  Health related quality of life (HRQoL) outcome
Score on the Whiteley Index | Within one year of screening
  Health anxiety outcome
Global brain volume | Within 2.5 years of screening
  Brain MRI measures
Segmental brain volume | Within 2.5 years of screening
  Brain MRI measures
Volume of white matter lesions | Within 2.5 years of screening
  Brain MRI measures
Number of clinical and subclinical infarcts | Within 2.5 years of screening
  Brain MRI measures
Number og micro-hemorrhages | Within 2.5 years of screening
  Brain MRI measures

CONTACTS AND LOCATIONS:
Overall Officials: Tor Ingenbrigtsen, Study Chair — University Hospital of North Norway
Locations (2):
- Norway (2):
  - Uit The Arctic University of Norway, Tromsø
  - University Hospital of North Norway Health Trust, Tromsø

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT07343895/Prot_000.pdf